CLINICAL TRIAL: NCT00474279
Title: Effects of an Oral GH Secretagogue (MK-677) on Body Composition and Functional Ability of Older Adults
Acronym: MOT089
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HIC #7444; NIH RO1 DK32632
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2007-05-16 (Estimated); Status verified 2007-05

CONDITIONS: Aging
Keywords: Growth hormone secretagogue; Body composition; Functional ability; Aging; Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — ibutamoren mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Orally active growth hormone secretagogue (MK-677)

SUMMARY:
The purpose of this study is to determine whether treatment of healthy older men and women with oral MK-677 for 12 months will enhance pulsatile GH release and increase mean GH and IGF-I concentrations into the range of young adults and will have favorable effects on body composition and functional ability on older adults.

DETAILED DESCRIPTION:
This is a two year, double-blind, placebo-controlled cross-over trial of once daily administration of MK-677, an oral GH secretagogue, to healthy older adults. During the first year, subjects will be randomized to MK-677 or placebo treatment. In each of three subgroups of subjects (men, women off and women on hormone replacement therapy), 16 subjects will receive MK-677 and 8 will receive placebo. After 1 year, the subjects who received placebo will be switched to MK-677 treatment; the subjects who received MK-677 for the first year will be randomized to either placebo or MK-677 for the second year of the study.The study will test changes in GH, IGF-I, body composition and function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women  60 years of age, with a body mass index of < 35 kg/m2.

Exclusion Criteria:

* Medication known to affect GH secretion, other than estrogen replacement therapy
* Coronary artery disease,
* Congestive heart failure,
* Peripheral vascular disease,
* Diabetes mellitus (requiring insulin or an oral hypoglycemic agent),
* Significant hypertension (BP >180 systolic or >100 diastolic at rest);
* Renal, hepatic, pulmonary disease;
* Untreated hypothyroidism, untreated hyperthyroidism;
* History of seizure disorder;
* History of malignancy (other than some skin cancers), history of active chronic infections (e.g., HIV, tuberculosis).
* Hematocrit < 40%, men, < 36%, women
* History of daily tobacco use within past 3 months
* Chronic alcohol abuse
* Strenuous exercise for average of more than 60 min/day
* Investigational drug within past 6 weeks
* Psychiatric history, especially anorexia nervosa
* Transmeridian travel within 2 weeks prior to or during study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 1998-07; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
At 12 months: 24-hour mean growth hormone concentrations
Insulin-like growth factor-I concentrations
Body weight and fat mass, specifically abdominal visceral fat
Fat-free mass
Safety determined by routine laboratory tests at 1 to 3 month intervals, yearly pap smears and mammograms

SECONDARY OUTCOMES:
at 12 months: Growth hormone secretory dynamics
Isokinetic muscle strength (knee and shoulder)
Thigh muscle cross-sectional area
Function tests (timed walks, stair climb, chair rise)
Quality of life assessments
Insulin sensitivity
Lipid profile
Resting metabolic rate
Aerobic exercise capacity
Exploratory outcomes:
effects of gender and HRT on primary outcomes
effects of treatment in year 2: Year 2 outcomes include effects of continuation on MK-677, or crossover to placebo, placebo to MK-677
bone mineral density at end of year 2.

CONTACTS AND LOCATIONS:
Overall Officials: Michael O. Thorner, MBBS, DSc,, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Chapman IM, Bach MA, Van Cauter E, Farmer M, Krupa D, Taylor AM, Schilling LM, Cole KY, Skiles EH, Pezzoli SS, Hartman ML, Veldhuis JD, Gormley GJ, Thorner MO. Stimulation of the growth hormone (GH)-insulin-like growth factor I axis by daily oral administration of a GH secretogogue (MK-677) in healthy elderly subjects. J Clin Endocrinol Metab. 1996 Dec;81(12):4249-57. doi: 10.1210/jcem.81.12.8954023.